CLINICAL TRIAL: NCT05503069
Title: Community Interventions to Improve Breastfeeding Rate in African American Mothers
Brief Title: Community Interventions to Improve Breastfeeding
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Norma Ojeda, Professor and Chair DABE, University of Mississippi Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Breastfeeding DN00486
Record Dates: First submitted 2022-08-01; First posted 2022-08-16 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Breastfeeding; Breastfeeding, Exclusive
Keywords: Breastfeeding; African American Mothers
MeSH Terms: conditions — Breast Feeding | interventions — Methods

STUDY DESIGN:
Intervention Model Description: This project will utilize a cohort case-controlled study design. There will be two arms with equally enrolled participants in each arm (1:1). Participants will be allocated in the control and intervention arm utilizing simple randomization with fixed number (n=60) for each arm distributed in group A (control) and group B (intervention). The participants will randomly select an envelope concealing the group label after signed the consent form.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - Control (No Intervention): The control group will receive standard of care, which include basic training by lactation educators.
- Group B - Intervention (Experimental): Women in the intervention arm will receive standard of care, which includes basic training in breastfeeding by lactation educators, and the action items related to the intervention.
  The intervention will include the following
  1. Providing a breast milk pumping machine to the mother,
  2. Facilitating training session to improve dietary literacy for lactating mothers,
  3. Distribution of educational material describing the benefits of continuing breastfeeding infants up to 12 months of age to family members, employers, day care managers/caregivers.
  Interventions: Behavioral: Interventions with social and cultural components

INTERVENTIONS:
Behavioral: Interventions with social and cultural components — Intervention Components
  * Enrollment: We are expecting an enrollment rate of 20 participants per week, and completing enrollment in 6 weeks (n=120 participants)
  * Baseline Data Collection
  * Distribution of Educational Materials
  * Lactation Training
  * Dietary Literacy Training
  * Follow Up Data collection: Infant's information on growth and development and Medical History of Infections, GI problems (diarrhea, constipation, colic, vomits, reflux) will be collected at 3, 6 and 12 months.
  * Follow UP Surveys: Mothers will complete a short survey at 3, 6, and 12 months exploring their breastfeeding behaviors and challenges.
  * Exit survey: Mothers will be asked to complete an exit survey on month 12 post-enrollment to explore their perception on the participation in the study.
  Arms: Group B - Intervention

SUMMARY:
The percentage of women breastfeeding their newborn babies is very low among minority populations such as African American women in Mississippi. There are good results with initiatives supporting the initiation of breastfeeding after delivery. However, the percentages of continuation of breastfeeding up to 3, 6 or 12 months are still very low in Mississippi. Therefore, this project is proposing to focus on community interventions including social and cultural components to promote and support continuation of breastfeeding.

* The social component will include interventions to promote supportive environments in the workplace for lactating mothers, as well as promoting the use of mother's milk to feed infants in daycare centers.
* The cultural component will focus on educating and raising awareness of the benefit of BF to prevent absenteeism at work, to reduce child illnesses, and to promote healthy child development. The cultural component will target the mother with her family and spouse/partner, employers, and daycare managers.

DETAILED DESCRIPTION:
The hypothesis of whether community interventions supporting breastfeeding practices will increase the rates of continuing breastfeeding at 6 and 12 months among African American women, will be tested with the following specific aims Aim 1: Will test whether providing breast milk pumping machine to lactating mothers will promote continuation of breastfeeding up to 6 and 12 months.

The intervention associated with this aim will include the provision of breast milk pumping machines free of charge to new mothers in the intervention arm at the time of discharge from the hospital. Mothers in the control group will follow standard of care practices, which do not include provision of pumping machines at discharge from the hospital.

Aim 2: Will test whether providing training to improve dietary literacy for lactating mothers will improve continuation of breastfeeding up to 6 and 12 months.

The intervention associated with this aim will include training session on topic related to dietary practices for lactating mothers.

Aim 3: Will test whether providing educational materials describing the benefits breastfeeding to family members, employers, and day care managers will improve continuing breastfeeding up to 6 and 12 months.

Study Design This project will utilize a cohort case-controlled study design. There will be two arms with equally enrolled participants in each arm (1:1). Participants will be allocated in the control and intervention arm utilizing simple randomization with fixed number (n=60) for each arm distributed in group A (control) and group B (intervention). The participants will randomly select an envelope concealing the group label after signed the consent form. The participants will open the envelope in front of research coordinator and the allocation group will be revealed.

The study will target African American women between 25 and 35 years of age who delivered singleton full term babies at the University of Mississippi Medical Center, without any perinatal complications. Babies of both sexes will be included. The Dyads of mother/infant participants will be randomized in the following groups: A- Control arm with n=60 participants, and B- Intervention arm with n=60 participants.

Women in the intervention arm will receive standard of care, which includes basic training in breastfeeding by lactation educators, and the action items related to the intervention.

The intervention will include the following

1. Providing a breast milk pumping machine to the mother,
2. Facilitating training session to improve dietary literacy for lactating mothers,
3. Distribution of educational material describing the benefits of continuing breastfeeding infants up to 12 months of age to family members, employers, day care managers/caregivers.

The control group will receive standard of care, which include basic training by lactation educators.

ELIGIBILITY:
Inclusion Criteria:

Women

* Age: 25 to 35 years of age
* Delivery: Full-term, singleton delivery at UMMC Infants
* Gestational Age: ≥ 37 weeks of gestation
* Sex: Both sexes

Exclusion Criteria:

Women

* Perinatal complication
* Medical indication to withhold breastfeeding practices Infants
* Prematurity
* Medical indication to withhold breastfeeding
* Congenital condition/malformation

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-25 (Estimated)

PRIMARY OUTCOMES:
Outcomes in Mothers at 3 months | At 3 months post enrollment.
  -Rates of continuation of breastfeeding at 3 months will be collected during the short phone interview.
Outcomes in Mothers at 6 months | At 6 months post enrollment.
  -Rates of continuation of breastfeeding at 6 months will be collected during the short phone interview.
Outcomes in Mothers at 12 months | At 12 months post enrollment.
  -Rates of continuation of breastfeeding at 12 months will be collected during the short phone interview.
Outcomes in Mothers Perceptions on Support at 12 months | At 12 months post enrollment.
  -Perception of mother on community support to promote breastfeeding will be explored with the exit survey.
Outcomes in Mothers Perceptions on Infant's wellbeing at 12 months | At 12 months post enrollment.
  -Perception of mother on infant wellbeing associated with breastfeeding practices will explored with exit survey.
Outcomes in Infant's development at 3 months | At 3 months post natal
  Development and growth using the percentile in growth chart will be collected at 3 months of age.
Outcomes in Infant's development at 6 months | At 6 months post natal
  Development and growth using the percentile in growth chart will be collected at 6 months of age.
Outcomes in Infant's development at 12 months | At 12 months post natal
  Development and growth using the percentile in growth chart will be collected at 12 months of age.
Outcomes in Infant's health at 3 months | At 3 months post natal
  -Incidence of infections and gastrointestinal problems will be collected at 3 months of age.
Outcomes in Infant's health at 6 months | At 6 months post natal
  -Incidence of infections and gastrointestinal problems will be collected at 6 months of age.
Outcomes in Infant's health at 12 months | At 12 months post natal
  -Incidence of infections and gastrointestinal problems will be collected at 12 months of age.

CONTACTS AND LOCATIONS:
Overall Officials: Norma B Ojeda, MD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center-Nursery Department of Pediatrics, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No
This study is not including a plan to share IPD with other researchers.

REFERENCES:
- [Background] O'Hare C, Kuh D, Hardy R. Association of Early-Life Factors With Life-Course Trajectories of Resting Heart Rate: More Than 6 Decades of Follow-up. JAMA Pediatr. 2018 Apr 2;172(4):e175525. doi: 10.1001/jamapediatrics.2017.5525. Epub 2018 Apr 2. PMID 29435577
- [Background] Schwarzenberg SJ, Georgieff MK; COMMITTEE ON NUTRITION. Advocacy for Improving Nutrition in the First 1000 Days to Support Childhood Development and Adult Health. Pediatrics. 2018 Feb;141(2):e20173716. doi: 10.1542/peds.2017-3716. Epub 2018 Jan 22. PMID 29358479
- [Background] Rantalainen V, Lahti J, Henriksson M, Kajantie E, Mikkonen M, Eriksson JG, Raikkonen K. Association between breastfeeding and better preserved cognitive ability in an elderly cohort of Finnish men. Psychol Med. 2018 Apr;48(6):939-951. doi: 10.1017/S0033291717002331. Epub 2017 Aug 22. PMID 28826414
- [Background] Indrio F, Martini S, Francavilla R, Corvaglia L, Cristofori F, Mastrolia SA, Neu J, Rautava S, Russo Spena G, Raimondi F, Loverro G. Epigenetic Matters: The Link between Early Nutrition, Microbiome, and Long-term Health Development. Front Pediatr. 2017 Aug 22;5:178. doi: 10.3389/fped.2017.00178. eCollection 2017. PMID 28879172
- [Background] Alakaam A, Lemacks J, Yadrick K, Connell C, Choi HW, Newman RG. Maternity Nurses' Knowledge and Practice of Breastfeeding in Mississippi. MCN Am J Matern Child Nurs. 2018 Jul/Aug;43(4):225-230. doi: 10.1097/NMC.0000000000000437. PMID 29958205
- [Background] Alakaam A, Lemacks J, Yadrick K, Connell C, Choi HW, Newman RG. Breastfeeding Practices and Barriers to Implementing the Ten Steps to Successful Breastfeeding in Mississippi Hospitals. J Hum Lact. 2018 May;34(2):322-330. doi: 10.1177/0890334417737294. Epub 2017 Nov 20. PMID 29156144
- [Background] Agostoni C, Marangoni F, Giovannini M, Galli C, Riva E. Prolonged breast-feeding (six months or more) and milk fat content at six months are associated with higher developmental scores at one year of age within a breast-fed population. Adv Exp Med Biol. 2001;501:137-41. doi: 10.1007/978-1-4615-1371-1_17. PMID 11787675